CLINICAL TRIAL: NCT03144999
Title: A Phase 1, Open-Label, Multi-Center, Dose-Escalating, Safety and Tolerability Study of a Single Intravitreal Injection of AAVCAGsCD59 in Patients With Advanced Non-Exudative (Dry) Age-Related Macular Degeneration With Geographic Atrophy
Brief Title: Treatment of Advanced Dry Age Related Macular Degeneration With AAVCAGsCD59
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: HMR-1001
Record Dates: First submitted 2017-05-02; First posted 2017-05-09 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Dry Age-related Macular Degeneration
Keywords: Dry AMD; Dry Age-related Macular Degeneration; Gene Therapy; Complement; Intravitreal Injection; Geographic Atrophy; Drusen; Membrane Attack Complex; CD59
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Intervention Model Description: This is a dose escalation study consisting of a low, mid, and high dose to evaluate the maximum tolerated dose (MTD). An additional 8 patients are enrolled at the MTD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose (Experimental): AAVCAGsCD59
  Interventions: Biological: AAVCAGsCD59
- Mid Dose (Experimental): AAVCAGsCD59
  Interventions: Biological: AAVCAGsCD59
- High Dose (Experimental): AAVCAGsCD59
  Interventions: Biological: AAVCAGsCD59

INTERVENTIONS:
Biological: AAVCAGsCD59 — AAVCAGsCD59 is administered as a single intravitreal injection in an office setting
  Other Names: HMR59

SUMMARY:
Age related macular degeneration (AMD) is the leading cause of vision loss in individuals over age 60. AMD is classified as wet and dry. Wet AMD constitutes 10 to 15% of all cases of AMD and occurs when an abnormal blood vessel grows in or under the retina leading to central vision loss. Wet AMD is successfully treated with injections in the eye on a monthly basis that stop the blood vessel from growing and leaking. The most common form of AMD is the dry variant or dry AMD that affects 85 to 90% of all patients with AMD. In dry AMD, there is loss of retinal pigment, formation of deposits called drusen, and loss of the vessels in a layer of the retina called the choriocapillaris. In the most severe forms of dry AMD there is loss of retinal tissue called geographic atrophy. Over time retinal tissue degenerates in the area responsible for central vision leading to vision loss leading to legal blindness. Currently no treatment for dry AMD exists so that there is a significant unmet need in patients with this ocular disease.

Recently, evidence has implicated an overactive inflammatory cascade called the complement system as playing a pivotal role in the development of dry AMD. The complement cascade consists of 3 arms that converge to form a pore-like complex on the surface of cells called the membrane attack complex (MAC). Accumulation of MAC on cell surfaces leads to cell damage and death causing the clinical findings seen in AMD. Normal cells within the human body produce a protein on their cell surfaces called CD59 that blocks the MAC from forming. In AMD, the complement cascade is upregulated and leads to more MAC formation than the body can protect itself against leading to cell destruction.

AAVCAGsCD59, an ocular gene therapy product that is injected in to the eye in the physician's office, causes normal retinal cells to increase the expression of a soluble form of CD59 (sCD59). This soluble recombinant version of the naturally occurring CD59 is designed and intended to protect retinal cells that are responsible for central vision by inhibiting the formation of the membrane attack complex (MAC), the terminal step of complement-mediated cell lysis. In gene therapy the cells of the retina are potentially permanently altered to make sCD59 for the life of the patient. With gene therapy only one injection is needed for the drug to be effective for the patient's entire life. This study will evaluate the safety after a single injection of AAVCAGsCD59 administered in an office setting for patients whose enrolled eye has advanced dry AMD with geographic atrophy. The initial study is 26 weeks followed by an additional 18-month safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 50 years of age or older
* Advanced dry AMD with GA in the study eye
* BCVA Snellen equivalent of 20/80 or worse in the study eye using ETDRS charts at a starting distance of 4m after the first 3 patients are enrolled and demonstrate favorable safety data
* Total GA lesion size 5mm2 (2 DA) to 20mm2 (8 DA) in the study eye; if multifocal, then at least one focus of GA needs to measure 1.27 mm2 (0.5 DA)
* Fellow eye BCVA of 20/800 or better and must be the eye with the better visual acuity
* Must be willing to undergo paracentesis of the anterior chamber

Exclusion Criteria:

* GA secondary to non AMD etiologies
* Prior or active choroidal neovascularization (CNV) in the study eye
* History of conditions in the study eye during screening which might alter visual acuity or interfere with study testing
* Active uncontrolled glaucoma
* Intraocular surgery in the study eye within 3 months of enrollment or are known or likely candidate for intraocular surgery (including cataract surgery) in the study eye within 1 year of treatment
* Acute or chronic infection in the study eye
* History of inflammation in the study eye or ongoing inflammation in either eye
* History of uveitis in the study eye
* Ongoing ocular inflammation in either eye
* Any contraindication to intravitreal injection
* Currently using or have used treatment for exudative AMD in the study eye only: laser photocoagulation, photodynamic therapy (PDT), ranibizumab (Lucentis®), pegaptanib sodium (Macugen®), bevacizumab (Avastin®) or aflibercept (Eylea®)
* Currently using any periocular (study eye), intravitreal (study eye) or systemic (oral or intravenous) corticosteroids within 3 months prior to screening.
* Any of the following underlying systemic diseases:

  * Unstable or severe cardiovascular disease, e.g., congestive heart failure (New York Heart Association Functional class III or IV), myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina, or critical limb ischemia;
  * Poorly controlled diabetes;
  * Clinically significant impaired renal or hepatic function, for example:
  * Cerebrovascular disease within 12 months prior to Screening;
  * Dementia or neurodegenerative disease (e.g., Alzheimer's disease, Parkinson's disease);
  * Have a malignancy at Screening or a history of malignancy that precludes completion of this 2-year study, including presence of tumor or disease whose treatment may directly affect the ability to evaluate the safety and efficacy of AAVCAGsCD59, or currently undergoing treatment for a specific cancer;
  * Immunocompromised conditions and/or need for immunosuppressive therapy;
* Any significant poorly controlled illness that would preclude study compliance and follow-up
* Current or prior use of any medication known to be toxic to the retina or optic nerve including, but not limited, to chloroquine/hydrochloroquine, deferoxamine, phenothiazines and ethambutol
* Previous treatment with any ocular or systemic gene transfer product
* Received any investigational product within 120 days prior to screening

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing ocular and systemic adverse events as graded by CTCAE v4.0 | 26 Weeks
  Measure intraocular inflammation, ocular changes and systemic side effects following a single intraocular injection of AAVCAGsCD59

SECONDARY OUTCOMES:
Evaluate the change in area of GA in eyes with dry AMD | 26 Weeks
  Efficacy of AAVCAGsCD59
Evaluate the rate of growth of GA in eyes with dry AMD | 26 Weeks
  Efficacy of AAVCAGsCD59
Incidence of conversion of dry AMD to wet AMD | 26 Weeks
  Efficacy of AAVCAGsCD59
Change in drusen volume measured by spectral domain OCT | 26 Weeks
  Efficacy of AAVCAGsCD59
Prevention of loss of 15 or more letters on an ETDRS visual acuity chart | 26 Weeks
  Efficacy of AAVCAGsCD59

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Heier, MD, Principal Investigator — Ophthalmic Consultants of Boston
Locations (1):
- Ophthalmic Consultants of Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No